CLINICAL TRIAL: NCT03429257
Title: Association Among Maternal Environmental Enteric Dysfunction, Aflatoxin Exposure, and Birth Outcomes: A Prospective Cohort Study in Mukono, Uganda
Brief Title: Maternal EED and Aflatoxin Birth Outcomes Study Uganda
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Shibani Ghosh, Adjunct Assistant Professor, Tufts University
Other Study IDs: AID-OAA-L-10-00006
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Birth Weight; Pregnancy Preterm; Aflatoxins Toxicity; Inflammatory Response
Keywords: Aflatoxin B1; Environmental Enteric Dysfunction; L:M Test; Pregnancy; Linear Growth Faltering; Birth Outcomes; Uganda
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples, Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women in Mukono Uganda: Single-group study
  Interventions: Other: Exposures of interest: Maternal EED and Aflatoxin Exposure

INTERVENTIONS:
Other: Exposures of interest: Maternal EED and Aflatoxin Exposure — Maternal EED, measured via lactulose: mannitol (L:M) ratios and serum concentrations of antibodies to the bacterial components flagellin and lipopolysaccharide (LPS); Maternal aflatoxin exposure, measured via serum concentration of AFB1-lysine adduct

SUMMARY:
This prospective cohort study focuses on the relationship between maternal environmental enteric dysfunction (EED) and maternal aflatoxin B1 exposure and birth outcomes, particularly infant anthropometry and gestational age, in Mukono, Uganda.

DETAILED DESCRIPTION:
The problem of stunting, which has long-term health and economic consequences both at the individual and population level, persists in low and middle income countries (LMICs). It has been recognized that an estimated 20% of stunting begins in-utero. Although poor maternal nutrition during pregnancy is often blamed, it has been hypothesized that maternal EED status and maternal aflatoxin exposure during pregnancy may also play a role. However, to date, there have been no studies which have attempted to show the association between EED in pregnant women and negative birth outcomes. Furthermore, few studies have examined the association between maternal aflatoxin exposure during pregnancy and negative birth outcomes.

In this prospective cohort study, pregnant women were enrolled at their first prenatal visit and birth outcome data was assessed within 48 hours of delivery. EED was measured via lactulose: mannitol (L:M) ratios and serum concentrations of antibodies to the bacterial components flagellin and lipopolysaccharide (LPS). Aflatoxin exposure was assessed by measuring the serum concentration of AFB1-lysine adduct from a blood sample taken at enrollment. Data on covariates were obtained from two surveys, one at enrollment and one three weeks prior to participant's estimated date of delivery.

The specific aims of this study were as follows:

1. To evaluate the relationship between markers of EED in pregnancy and negative birth outcomes, including low birth weight, stunting at birth, small head circumference, and premature delivery.
2. To evaluate the relationship aflatoxin B1 exposure in pregnancy and negative birth outcomes, including low birth weight, stunting at birth, small head circumference, and premature delivery.

ELIGIBILITY:
Inclusion Criteria:

* Carrying a singleton pregnancy
* 18-45 years old
* Residing within 10 kilometers of Mukono Town

Exclusion Criteria:

* Younger than 18 years old or older than 45 years old
* HIV-positive (verified via routine rapid HIV test conducted at first prenatal visit)
* Severely malnourished (defined as BMI <16.0 kg/m^2)
* Severely anemic (defined as Hb <7 g/dl)
* Planning to move away from Mukono District prior to delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women aged 18-45 years who visited Mukono Health Center IV in Mukono, Uganda for their first prenatal visit and who qualified for the study based on inclusion/exclusion criteria were invited to join the study until enrollment target was met.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Infant Birth Weight | Measured within 48 hours of delivery
  Low birth weight < 2500 grams
Infant Birth Length | Measured within 48 hours of delivery
Infant Gestational Age at Birth | Measured within 48 hours of delivery
  Preterm birth <37 weeks gestation
Infant Head Circumference | Measured within 48 hours of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Shibani Ghosh, PhD, Principal Investigator — Tufts University Friedman School of Nutrition Science and Policy
Locations (1):
- Mukono Health Center IV, Mukono, Uganda

IPD SHARING:
Plan to Share IPD: No